CLINICAL TRIAL: NCT05136001
Title: Characterizations of Gut Microbiota and Postoperative Sleep in Patients Undergoing Heart Valve Surgery With Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Professor, China Medical University, China
Other Study IDs: 2021.09.10-02
Record Dates: First submitted 2021-11-06; First posted 2021-11-26 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Heart Valve Surgery
Keywords: Gut Microbiota; polysomnography
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — gut microbiota and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: polysomnography — Duration of sleep was collected with polysomnography on second postoperative night. (from 20:00pm to 06:00am).

SUMMARY:
The investigators designed a study to assess whether there is any change in gut microbiota and postoperative sleep before and after heart valve surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
The investigators designed a study to assess whether there is any change in gut microbiota and postoperative sleep before and after heart valve surgery with cardiopulmonary bypass. Firstly, this study aims to characterize the gut microbiota in patients with valve disease treated with surgery. Secondly, it aims to evaluate microbiota and its influence on postoperative sleep.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese;
* Age, 18 to 65 years old;
* Patients undergoing heart valve surgery with cardiopulmonary bypass

Exclusion Criteria:

* Preoperative Pittsburgh Sleep Quality Index global scores higher than 6
* Cognitive difficulties
* Partial or complete gastrectomy
* Previous esophageal surgery
* Previous treated by radiotherapy or surgery
* Inability to conform to the study's requirements
* Body mass index exceeding 30 kg/m2
* Deprivation of a right to decide by an administrative or juridical entity
* Ongoing participation or participation in another study <1 month ago
* Recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or traditional Chinese medicine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will characterize the gut microbiota and serum metabolites in one group of 36 patients before and after heart valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
gut microbiota | from baseline to postoperative 72 hours
  This study will characterize the gut microbiota in one group of 36 patients before and after heart valve surgery

SECONDARY OUTCOMES:
postoperative sleep | on the second postoperative night from 20:00 to 6:00
  This study will characterize the postoperative sleep measured by polysomnography in one group of 36 patients after heart valve surgery
serum metabolites | from baseline to postoperative 72 hours
  This study will characterize the serum metabolites in one group of 36 patients before and after heart valve surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided